CLINICAL TRIAL: NCT05849129
Title: Adjunctive Intravenous Ascorbic Acid for Advanced Non-Small Cell Lung Cancer: A Double Blind, Placebo Controlled, Phase II Randomized Controlled Trial
Brief Title: Adjunctive Intravenous Ascorbic Acid for Advanced Non-Small Cell Lung Cancer
Acronym: AIVAA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Ottawa Hospital Research Institiute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20220721-01H
Record Dates: First submitted 2023-04-24; First posted 2023-05-08 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Ascorbic Acid; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Vitamin C (Experimental): 1g/kg IVC administered twice weekly for 6 months.
  Interventions: Drug: Ascorbic acid
- Normal Saline (Placebo Comparator): Equivalent volume normal saline administered twice weekly for 6 months.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Ascorbic acid — High dose ascorbic acid delivered intravenously
  Other Names: Vitamin C
  Arms: Intravenous Vitamin C
Other: Normal Saline — 0.9% NaCl solution
  Other Names: Sodium Chloride Solution
  Arms: Normal Saline

SUMMARY:
This is a two arm RCT evaluating the effect of intravenous vitamin C versus placebo in patients with incurable non-small cell lung cancer. Participants in both arms will be receiving platinum doublet chemotherapy with or without concurrent immunotherapy as standard care. We plan to enroll 90 patients over 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years of age) seen at TOHCC with stage IIIB or IV primary non-small cell lung cancer
2. Eligible and scheduled for first line platinum-doublet chemotherapy with or without concurrent immunotherapy

Exclusion Criteria:

1. ECOG status greater than 2
2. Previously received IVC within 6 months prior to randomization
3. Biochemical deficiency in G6PD
4. Estimated Glomerular Filtration Rate (eGFR) less than 45 mL/min
5. Currently taking insulin or warfarin
6. History of severe renal dysfunction or hemochromatosis
7. Previously undergone cytotoxic chemotherapy or immunotherapy within 12 months prior to randomization
8. If pregnant or planning to become pregnant: not a carrier of the gene for G6PD deficiency
9. Currently taking an investigational product or participation in an investigational study within the past 30 days
10. Any reason which, under the discretion of the Principal Investigator or delegate, would preclude the patient from participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2030-10-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life | Baseline, Chemo cycles 1-4, 6 months, 12 months
  Participant reported quality of life (QOL) measured using the Functional Assessment of Cancer Therapy - Lung (FACT-L). FACT-L is a validated tool for assessing QOL in patients with lung cancer. FACT scores are normalized to values between 0-100, where 0 is the worst QOL and 100 is the best QOL imaginable. Each chemotherapy cycle is 3 weeks in length.

SECONDARY OUTCOMES:
Chemotherapy-Related Toxicities | 12 months
  Frequency of adverse events (AE) which are commonly experienced by patients undergoing chemotherapy. Measured using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE). 31 symptoms were selected by the investigators.
Frequency of Discontinuation of Chemotherapy | 6 months
  Patients often discontinue chemotherapy due to side effects. The investigators will monitor the incidence of stopping chemotherapy and compare the number of patients who stop chemotherapy in both arms.
Change in General Symptom Burden | Baseline, chemo cycles 1-4, 6 months, 12 months
  Measured using the Edmonton Symptom Assessment Scale, which measures 9 symptoms commonly experienced by cancer patients. Each symptom is rated on a scale of 0-10, where 0 is the best symptom and 10 is the worst symptom. Each chemotherapy cycle is 3 weeks in length.
Change in C-Reactive Protein Levels | Baseline, chemo cycles 1-4, 6 months, 12 months
  The investigators will monitor the changes in C-reactive protein (CRP), a common indicator of systemic inflammation. Mean changes in CRP will be compared between arms. Each chemotherapy cycle is 3 weeks in length.
Tumour Progression | 12 months
  The investigators will monitor tumour progression using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, which measures the incidence of complete response, partial response, stable disease, and progressive disease during treatments.
Survival | 24 months
  The incidence of all cause mortality will be compared between arms.
Safety | 6 months
  The investigators will monitor the incidence of all adverse events in both arms to add to the safety profile of IVC in this population.
Cytotoxicity | 12 months
  The investigators will assess the ability of IVC to bring serum ascorbate levels to at least 15mM, which is the hypothesized level at which cytotoxic effects may occur. Levels 15mM or above will be considered adequate.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. Cumulative data not present in the manuscript or on this website may be shared upon request.